CLINICAL TRIAL: NCT07315048
Title: Application of Healthcare Failure Mode and Effect Analysis in Nursing Risk Management of Emergency Surgery for Patients With Spontaneous Subarachnoid Hemorrhage
Brief Title: Nursing Risk Management in Emergency SAH Surgery Using Healthcare Failure Mode and Effect Analysis(HFMEA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Lan, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: WestChinaH-HX-2025-04
Record Dates: First submitted 2025-12-08; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Spontaneous Subarachnoid Hemorrhage
Keywords: Healthcare Failure Mode and Effect Analysis; Nursing Risk Management; Emergency Surgery; Patient Safety
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients assigned to the intervention arm received every element of conventional emergency neurosurgical care plus a structured, prospective safety overlay derived from Healthcare Failure Mode and Effect Analysis. The add-on programme was delivered by a nine-member, hospital-authorised HFMEA team (one chief neurosurgeon, two attending neurosurgeons, one head nurse, four bedside nurses, one quality-manager) who had completed an 8-hour training course on HFMEA principles, risk-priority-number (RPN) scoring and decision-tree analysis. The programme ran from the minute the participant arrived in the emergency department until 30-days post-operation and consisted of six sequential steps that were re-applied every month.
  Interventions: Behavioral: HFMEA-based nursing-risk programme
- Control group (No Intervention): The control group received conventional nursing risk management, including:
  1. Admission assessment: vital signs monitoring, neurological function assessment, Hunt-Hess grading;
  2. Preoperative nursing: condition observation, psychological care, preoperative preparation;
  3. Postoperative nursing: close monitoring of vital signs, neurological function observation, complication prevention;
  4. Health education: disease knowledge, precautions, rehabilitation guidance;
  5. Discharge guidance: medication instructions, follow-up arrangements, lifestyle recommendations.

INTERVENTIONS:
Behavioral: HFMEA-based nursing-risk programme — Alongside standard care, these patients were managed with an HFMEA-based safety bundle. A trained nine-member team had pre-identified 12 highest-risk failure points (delayed ICP checks, missed re-bleeding signs, vasospasm, seizures, infection, etc.). From admission to day-30, nurses followed printed checklists and electronic order-sets: neuro-vitals every 15-30 min, BP target 140-160 mmHg, daily TCDs, automatic "red-flag" escalation for sudden headache/GCS drop, Triple-H protocol for velocities >120 cm/s, prophylactic levetiracetam for severe grades, 30° head positioning, chlorhexidine/line bundles, pain-delirium scale, bed-alarm, SBAR hand-over and a 5-minute family video with teach-back. Compliance was tracked in real time and reviewed monthly; measures were updated if failure rates did not fall within six weeks.
  Arms: Intervention group

SUMMARY:
The investigators are testing whether a new nurse-led safety program (HFMEA) lowers problems during emergency brain-aneurysm surgery better than usual care.

Adults with a sudden brain bleed (subarachnoid hemorrhage) who need urgent clipping or coil placement at the hospital are randomly placed in one of two groups:

Usual nursing care, or Usual care plus HFMEA (nurses use checklists to spot and prevent risks such as re-bleeding, high brain pressure, infection, seizures).

The investigators count how often any nursing-related problems happen within 30 days after surgery, how long patients stay, and how satisfied the participants and their families are.

Results will show if this extra safety program should become standard practice.

DETAILED DESCRIPTION:
A single-center randomized trial of adults patients undergoing emergency repair for ruptured brain aneurysms was trying to determing that if proactive "Healthcare Failure Mode and Effect Analysis" (HFMEA) could lower the rate of nursing-related adverse events from 1 in 5 patients to fewer than 1 in 15.

Nurses trained in HFMEA mapped every step of care-from arrival through discharge-identified the 12 highest-risk moments (e.g., delayed pressure checks, missed re-bleeding signs), and built checklists, alert thresholds, and team huddles to stop problems before they started.

aim: adding a structured, forward-looking safety drill to routine neuro-critical nursing appears to spare two out of every three avoidable complications after emergency "brain-aneurysm" surgery without extra technology or cost.

ELIGIBILITY:
Inclusion Criteria:

1. sSAH confirmed by head CT and/or CT angiography (CTA) or digital subtraction angiography (DSA), with identified intracranial aneurysm;
2. Age 18-75 years;
3. Time from onset to admission ≤72 hours;
4. Undergoing emergency surgical treatment (open aneurysm clipping or endovascular coiling);
5. Hunt-Hess grade I-V;
6. Patient or family consent to participate in the study with signed informed consent.

Exclusion Criteria:

1. Traumatic subarachnoid hemorrhage;
2. Concurrent other intracranial diseases (e.g., brain tumors, arteriovenous malformations);
3. Severe cardiac, hepatic, or renal dysfunction;
4. Coagulation disorders;
5. History of psychiatric disorders or cognitive impairment;
6. Pregnancy or lactation;
7. Transfer to another hospital or treatment withdrawal.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
perioperative nursing adverse event | 30 days
  Incidence of perioperative nursing adverse events, including:
  * Rebleeding
  * Cerebral vasospasm
  * Increased intracranial pressure
  * Seizures
  * Pulmonary infection
  * Pressure ulcers
  * Deep vein thrombosis
  * Catheter-related infections
  * Falls/bed exits
  * Medication errors, etc.

SECONDARY OUTCOMES:
Nursing Quality Score | 30 days
  Nursing Quality Score: Newcastle Satisfaction with Nursing Scale (NSNS), including four dimensions: condition observation, basic nursing, specialized nursing, and health education, each scored 0-25 points, total score 0-100 points, with higher scores indicating better nursing quality.
Patient Satisfaction Score | 30 days
  Self-designed satisfaction questionnaire covering nursing attitude, nursing skills, health education, environmental management, using 5-point Likert scale, total score 20-100 points.
Family Satisfaction Degree | 30 days
  Family satisfaction questionnaire assessing overall satisfaction with nursing services.
Length of Hospital Stay | 30 days
  Days from admission to discharge.
30-day Mortality | 30 days
  All-cause mortality within 30 days postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol